CLINICAL TRIAL: NCT06171984
Title: Thrombophilia Assessment Under Direct Oral Anticoagulants (DOAC): Efficacy of Activated Charcoal
Brief Title: Thrombophilia Assessment Under DOAC: Effectiveness of Activated Charcoal
Acronym: DOAC-Stop
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8673
Record Dates: First submitted 2022-09-06; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Thrombophilia
Keywords: Thrombophilia; direct oral anticoagulants; DOAC; Apixaban; Rivaroxaban; Dabigatran; Hemostasis tests
MeSH Terms: conditions — Thrombophilia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Direct oral anticoagulants (DOAC) are anticoagulant molecules that act either directly on factor Xa (Apixaban, Rivaroxaban) or on factor IIa (Dabigatran).

AODs interfere with most coagulation tests, especially those performed by chronometric technique.

For this reason, part of the thrombophilia workup (protein S, search for lupus anticoagulants, antithrombin for patients on dabigatran) cannot be performed on DOACs at the HUS.

Recent studies have highlighted the effectiveness of activated charcoal to adsorb DOACs in order to perform certain hemostasis tests.

ELIGIBILITY:
Inclusion criteria:

* Adult subject (≥ 18 years of age)
* Blood sample already analyzed in a usual way in the laboratory as part of the care
* Subject not objecting to the reuse of his or her medical data for scientific research purposes.

Exclusion criteria:

- Insufficient sample

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult subject (≥ 18 years of age) with blood sample already analyzed in a usual way in the laboratory of HUS as part of the care
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01-19 (Estimated)

PRIMARY OUTCOMES:
Interference or not of activated charcoal in the measurement of protein S, antithrombin, and in the search for lupus anticoagulants. | Through study completion, an average of 6 months
  This study compares the results of two diagnostic techniques (Thrombophilia work-up under direct oral anticoagulants (DOACs)), one using activated charcoal versus another not using it

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratoire d'Hématologie - CHU de Strasbourg - France, Strasbourg, France